CLINICAL TRIAL: NCT02076399
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Study of Fostamatinib Disodium in the Treatment of Persistent/Chronic Immune Thrombocytopenic Purpura
Brief Title: A Efficacy and Safety Study of R935788 in the Treatment of Persistent/Chronic Immune Thrombocytopenic Purpura (ITP)
Acronym: FIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-935788-047; 2013-005452-15 (EudraCT Number)
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2018-10

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Persistent Immune Thrombocytopenic Purpura; Chronic Immune Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fostamatinib Disodium (Experimental): Subjects begin with Fostamatinib Disodium tablet 100 mg PO bid and increase to 150 mg big after week 4 based on platelet count and tolerability.
  Interventions: Drug: Fostamatinib disodium
- Placebo (Other): Placebo tablet PO bid (morning and evening) over the course of 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fostamatinib disodium — Fostamatinib (100 mg PO bid or 150 mg PO bid)
  Other Names: R935788; R788; Fostamatinib
  Arms: Fostamatinib Disodium
Drug: Placebo — Placebo tablet PO bid (morning and evening) over the course of 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether fostamatinib is safe and effective in the treatment of persistent/chronic Immune Thrombocytopenic Purpura (ITP).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of persistent/chronic ITP for at least 3 months.
* Average platelet count < 30,000/µL (and none > 35,000 unless as a result of rescue therapy) from at least 3 qualifying counts

Exclusion Criteria:

* Clinical diagnosis of autoimmune hemolytic anemia
* Uncontrolled or poorly controlled hypertension
* History of coagulopathy including prothrombotic conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-07-14 (Actual); Primary Completion 2016-04-21 (Actual); Study Completion 2016-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rigel Pharmaceuticals, Inc., Study Director — Rigel Pharmaceuticals,Inc.
Locations (52):
- United States (13):
  - Arizona Oncology Associates, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Bleeding & Clotting Disorders Institute, Peoria, Illinois
  - Horizon Oncology Research, Inc, Lafayette, Indiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - Bill Hefner VA Medical Center, Salisbury, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Signal Point Clinical Research Center LLC, Middletown, Ohio
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
- Australia (9):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Launceston General Hospital, Launceston, Tasmania
  - Frankston Hospital, Frankston, Victoria
  - Dept of Haematology, The Alfred Hospital and Monash Medical Centre, Melbourne, Victoria
  - Perth Blood Institute, Nedlands, Western Australia
- Canada (3):
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- Denmark (4):
  - Herlev Hospital University of Copenhagen, Department of Hematology L124, Herlev, DK
  - Dept. of Haematology, Odense University Hospital, Odense C, DK
  - Hematological department, Roskilde Hospital, Roskilde, DK
  - Aarhus University Hospital, Aalborg
- Hungary (3):
  - Semmelweis University 1st, Budapest
  - University of Debrecen, Debrecen
  - Pecs University, Pécs
- Italy (5):
  - Ematologia - Padigilione 8, Policinico S. Orsola Malpighi, Azienda Ospedaliero Universitaria di Bologna, Bologna
  - Ospedale San Raffaele S.r.l. Dipartimento di Oncoematologia, Milan
  - Universitã Federico II di Napoli, Napoli
  - OspedaleCivile-ClinicaEmatologica/PUGD, Udine
  - ULSS 6 Vicenza-Ospedale San Bortolo di Vicenza, Vicenza
- HAGA ziekenhuis, Haag, NL, Netherlands
- United Kingdom (14):
  - Kent & Canterbury Hospital, Kent, Canterbury
  - Colchester General Hospital, Colchester, Essex
  - Royal Liverpool University Hospital, Liverpool, UK
  - St. James's Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Royal London Hospital, London
  - Hammersmith Hospital, Catherine Lewis Centre, London
  - University College Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - James Paget University Hospital, Norfolk
  - Oxford University Hospital, Oxford
  - University Hospital of North Staffordshire, Stoke-on-Trent
  - Sandwell General Hospital, West Bromwich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cooper N, Altomare I, Thomas MR, Nicolson PLR, Watson SP, Markovtsov V, Todd LK, Masuda E, Bussel JB. Assessment of thrombotic risk during long-term treatment of immune thrombocytopenia with fostamatinib. Ther Adv Hematol. 2021 Apr 30;12:20406207211010875. doi: 10.1177/20406207211010875. eCollection 2021. PMID 33995988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 76 patients were enrolled from July 2014 to April 2016
Groups:
- Fostamatinib Recipient: Fostamatinib (100 mg PO bid or 150 mg PO bid)
- Placebo Recipient: Placebo
Period: Overall Study
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Started | 51 | 25
Completed | 12 | 1
Not Completed | 39 | 24

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Fostamatinib Recipient | Placebo Recipient | Total
Number analyzed (Participants) | 51 | 25 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (17.7) | 53.2 (16.0) | 56.0 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 17 | 47
  Male | 21 | 8 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 48 | 24 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 44 | 21 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stable Platelet Response (Count of ≥50,000/µL on at Least 4 of the Last 6 Scheduled Visits Between Weeks 14 and 24)
Description: A stable platelet response by Week 24 defined as a platelet count of at least 50,000/μL on at least 4 of the last 6 scheduled visits between Weeks 14 and 24
Time Frame: From Week 14 to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 51 | 25
Participants | 9 | 0
Statistical Analysis 1: Comparison: Fostamatinib Recipient vs Placebo Recipient; Test type: Superiority; p = 0.0261, Fisher Exact; Risk Difference (RD) = 17.6, 95% CI 2-sided [7.2 to 28.1]

2. Secondary Outcome: Number of Participants With Platelet Count ≥ 50,000/µL at Week 12
Description: Platelet Count ≥ 50,000/µL at Week 12
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 51 | 25
Participants | 11 | 0

3. Secondary Outcome: Number of Participants With Platelet Count ≥ 50,000/µL at Week 24
Description: Platelet Count ≥ 50,000/µL at Week 24
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 51 | 25
Participants | 8 | 0

4. Secondary Outcome: Platelet Count ≥ 30,000/μL and ≥ 20,000/μL Above Baseline in Subjects With Baseline Platelet Count of <15,000/μL at Week 12.
Description: Number of subjects with baseline platelet count <15,000/μL who showed platelet count increase to ≥30,000/μL and ≥20,000/μL from baseline count at Week 12.
Time Frame: Baseline to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 25 | 12
Participants | 4 | 0

5. Secondary Outcome: Platelet Count ≥ 30,000/μL and ≥ 20,000/μL Above Baseline in Subjects With Baseline Platelet Count of <15,000/μL at Week 24.
Description: Number of subjects with baseline platelet count <15,000/μL who showed platelet count increase to ≥30,000/μL and ≥20,000/μL from baseline count at Week 24.
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 25 | 12
Participants | 4 | 0

6. Secondary Outcome: Mean of the ITP Bleeding Score (IBLS)
Description: The ITP Bleeding Scale (IBLS) is an immune thrombocytopenic purpura (ITP)-specific bleeding score used to analyze the correlation of clinical and laboratory platelet variables with bleeding. The IBLS comprises of 11 grades from 0 (none) to 2 (marked bleeding) by history over the previous week or by exam; 2 being worse. These 11 grades include: skin by physical exam, oral by physical exam, skin by history, oral by history, epistaxis, gastrointestinal, urinary, gynecological, pulmonary, intracranial hemorrhage, and subconjunctival hemorrhage. After each grade is scored, the mean value for all 11 grades is calculated (lowest score being 0 and highest score being 2) for each subject visit. LOCF method was used to impute any missing data.
  The mean of the IBLS scores across visits during the 24-week treatment period was summarized by treatment group using descriptive statistics. A 2-sided, 2-sample t-test was used to test for a difference in means between treatments for this endpoint.
Time Frame: Assessed over the 24-week study period
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 51 | 25
scores on a scale | 0.13 (0.12) | 0.14 (0.10)
Statistical Analysis 1: Comparison: Fostamatinib Recipient vs Placebo Recipient; Test type: Superiority; p = 0.6642, t-test, 2 sided — P-value from a two-sided two-sample t-test, testing for a difference in means between fostamatinib and placebo; Risk Difference (RD) = -0.01, 95% CI 2-sided [-0.01 to 0.0]

7. Secondary Outcome: Mean of World Health Organization (WHO) Bleeding Scale
Description: The World Health Organization (WHO) bleeding scale is a standardized grading scale created to measure the severity of bleeding. The scale is a clinical investigator-assessed five-point scale with a score range starting at the lowest 0=No bleeding, 1 = Petechiae, 2=Mild blood loss, 3=Gross blood loss, to the worse 4=Debilitating blood loss. The WHO bleeding scale is scored by history over the previous-week or by exam. After each grade is scored, the mean value is calculated (lowest score being 0 [no bleeding] to the highest score being 4 [debilitating blood loss]) for each visit. LOCF method was used to impute any missing data.
  The mean of the WHO bleeding scale across visits during the 24-week treatment period was summarized by treatment group using descriptive statistics. A 2-sided, 2-sample t-test was used to test for a difference in means between treatments for this endpoint.
Time Frame: Assessed over the 24-week study period
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Fostamatinib Recipient | Placebo Recipient
Number analyzed (Participants) | 51 | 25
scores on a scale | 0.61 (0.66) | 0.46 (0.56)
Statistical Analysis 1: Comparison: Fostamatinib Recipient vs Placebo Recipient; Test type: Superiority; p = 0.3365, t-test, 2 sided — P-value from a two-sided two-sample t-test, testing for a difference in means between fostamatinib and placebo; Risk Difference (RD) = 0.15, 95% CI 2-sided [-0.2 to 0.5]

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | Fostamatinib Recipient | Placebo Recipient
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/25
Serious Adverse Events (participants affected / at risk) | 8/51 | 5/25
Other Adverse Events (participants affected / at risk) | 49/51 | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostamatinib Recipient (N=51) | Placebo Recipient (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Retinal Tear (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fostamatinib Recipient (N=51) | Placebo Recipient (N=25)
Diarrhoea (Gastrointestinal disorders) | 21 | 4
Nausea (Gastrointestinal disorders) | 15 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Alanine aminotransferase increased (Investigations) | 9 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 0
Blood pressure increased (Investigations) | 3 | 1
Headache (Nervous system disorders) | 7 | 6
Dizziness (Nervous system disorders) | 9 | 4
Dysgeusia (Nervous system disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Fatigue (General disorders) | 6 | 1
Pyrexia (General disorders) | 2 | 2
Chest pain (General disorders) | 4 | 1
Hypertension (Vascular disorders) | 13 | 1
Rash (Vascular disorders) | 4 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No